CLINICAL TRIAL: NCT02146066
Title: An Expanded Access Protocol for the Treatment of Glioblastoma Multiforme in Patients With Already Manufactured DCVax®-L, Autologous Dendritic Cells Pulsed With Tumor Lysate Antigen Who Have Screen-Failed Protocol 020221
Brief Title: Expanded Access Protocol for GBM Patients With Already Manufactured DCVax®-L Who Have Screen-Failed Protocol 020221
Acronym: DCVax-L EAP
Status: Available | Type: Expanded Access
Sponsor: Northwest Biotherapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: 0202EA
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: GBM; Glioblastoma Multiforme
Keywords: GBM; Brain tumor; glioblastoma; Brain tumor WHO grade IV
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

INTERVENTIONS:
Biological: DCVax-L — Autologous Dendritic Cells Pulsed with Tumor Lysate Antigen

SUMMARY:
The study is an open-label expanded access study for patients for whom vaccine was manufactured during the Northwest Biotherapeutics' 020221 DCVax-L for GBM screening process, but who subsequently failed to meet specific enrollment criteria. Patients will receive therapy per investigator discretion (standard of care) as well as active vaccine per the 020221 protocol administration schedule. It is estimated that approximately 99 patients will enroll in this study.

DETAILED DESCRIPTION:
Patients who are being screened under protocol 020221 who are not eligible for enrollment due to a) evidence of disease progression or pseudo-progression post chemo-radiation or b) insufficient (<5 doses) vaccine manufactured, and for whom the DCVax-L treatment was manufactured and released are eligible for this study.

Treatment Schedule:

Open label vaccine injections will be give per the associated 020221 protocol. Injections will be given at days 0, 10, 20, and at months 2, 4, 8, 12, 18, 24 and 30. There are no therapeutic restrictions, but guidelines for drug administration are recommended as per the 020221 protocol.

Data collected includes vaccine administration information, and any vaccine related adverse event. Patient MRIs will be collected centrally for future review. Patients will be followed for disease progression and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Screen-Fail for protocol 020221 due to either:

   * Radiographic evidence of disease progression or pseudoprogression at the Baseline visit under protocol 020221, as determined by central imaging review, OR
   * Insufficient vaccine manufactured for protocol 020221 (i.e. less than 5 doses).
2. Patients must have a KPS rating of ≥70 at the Baseline Visit (Visit 5) (refer to Appendix D, Performance Status Scales).
3. Patients may have received steroid therapy as part of their primary treatment. Steroid treatment should preferably be stopped; or if continued steroid use is clinically indicated, be tapered down to no more than 4 mg dexamethasone qd at least 7 days prior to the first immunization .
4. DCVax-L product manufactured and released.

Exclusion Criteria:

1. Active uncontrolled infection, or acute infection requiring antibiotic or antifungal therapy. Antibiotic and antifungal therapy should be completed approximately 7 days prior to the first immunization.
2. Fever ≥101.5oF. If considered possibly transient, retesting is allowed.
3. Unstable or severe intercurrent medical conditions.
4. Females of child-bearing potential who are pregnant or lactating or who are not using adequate contraception (abstinence, surgical, hormonal or double barrier, i.e. condom and diaphragm). 020221 Baseline lab results and or local lab results are acceptable.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCLA Medical Center, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - St. Joseph Hospital of Orange, Orange, California
  - University of California, Irvine Medical Center, Orange, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Colorado Neurological Institute, Englewood, Colorado
  - University of Florida, Gainesville, Florida
  - Memorial Healthcare System Memorial Cancer Institute, Hollywood, Florida
  - Cadence Cancer Center at Warrenville, Warrenville, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - John Nasseff Neuroscience Institute - Abott Northwestern Hospital, Minneapolis, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Capital Health, Trenton, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Columbia University Medical Center Neurological Institute of New York, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Saint Thomas Research Institute, Nashville, Tennessee
  - Swedish Neuroscience Institute, Seattle, Washington
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin